CLINICAL TRIAL: NCT02273349
Title: Evaluation of the PneumRx, Inc. Lung Volume Reduction Coil for the Treatment of Emphysema in Alpha-1 Antitrypsin Deficient Patients
Brief Title: Lung Volume Reduction Coils for Emphysema in Alpha-1 Antitrypsin Deficiency
Acronym: LuReCAA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL001-AATD
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Alpha-1-Antitrypsin Deficiency; Chronic Obstructive Lung Disease; Emphysema
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Patients with Alpha-1-Antitrypsin deficiency treated with endoscopic lung volume reduction using Lung Volume Reduction Coils (PneumRx Inc.)
  Interventions: Device: Lung Volume Reduction Coil (PneumrX Inc.)

INTERVENTIONS:
Device: Lung Volume Reduction Coil (PneumrX Inc.) — Endoscopic Lung Volume Reduction

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the RePneu Lung Volume Reduction Coil (LVRC) in patients with Alpha-1-Antitrypsin deficiency (AATD) caused emphysema. The hypothesis is that emphysema in AATD patients shows similar tissue destruction profile was well as symptoms and thus will respond favorably to LVRC treatment, demonstrating improvement in lung function, exercise capacity, and quality of life relative to their baseline status.

ELIGIBILITY:
Inclusion Criteria:

1. Patient > 18 years of age, diagnosed with AATD emphysema
2. CT scan indicates bilateral heterogeneous or non-severe homogeneous emphysema, with sufficient lung parenchyma for coil deployment, in accordance with manufacturer recommendations (see section 5.2.4.1).
3. Patient has post- bronchodilator FEV1 less than or equal to 45% predicted
4. Total Lung Capacity > 100%
5. Residual Volume (RV) >175% predicted
6. Patient has stopped smoking for a minimum of 8 weeks prior to entering the study
7. Patient has read, understood and signed the Informed Consent form
8. Patient is willing and able to attend all required follow-up visits
9. Patient is willing and able to undergo bilateral LVRC treatment
10. Patient has received Pneumococcal and Influenza vaccinations consistent with local recommendations and/or policy

Exclusion Criteria:

1. Patient has a change in FEV1 > 20% post-bronchodilator.
2. Patients DLCO < 20% predicted
3. Patient has a history of recurrent clinically significant respiratory infection
4. Patient has uncontrolled pulmonary hypertension defined by right ventricular pressure >50mmHg and or evidenced by echocardiogram
5. Patient has an inability to walk >140 meters (150 yards) in 6 minutes
6. Patient has evidence of other disease that may compromise survival such as lung cancer, renal failure, etc.
7. Patient is pregnant or lactating
8. Patient has an inability to tolerate bronchoscopy under moderate sedation or anesthesia
9. Patient has clinically significant bronchiectasis
10. Patient has giant bullae > 1/3 lung volume
11. Patient has had previous LVR surgery, lung transplant or lobectomy
12. Patient has been involved in other pulmonary drug or device studies with 30 days prior to this study
13. Patient is taking > 20mg prednisone (or similar steroid) daily
14. Patient is on an antiplatelet agent (such as Plavix) or anticoagulant therapy (such as heparin or coumadin) or has not been weaned off prior to procedure
15. Patient has other condition that would interfere with completion of study, follow up assessments or that would adversely affect outcomes
16. Patient has severe homogeneous emphysema by CT scan.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
symptomatic improvement in St. George's Respiratory Questionnaire (SGRQ) from Baseline (Pre-Treatment Visit) compared to the 6 months Follow-up Visit | 6 months
  Quality of Life

SECONDARY OUTCOMES:
Percent change in FEV1 from Baseline (Pre-Treatment Visit) | 6 and 12 months
  Lung function
Decrease in the Residual Volume and the RV/TLC ratio | 6 and 12 months
  Lung function
Improvement in the 6 minute walk distance | 6 and 12 months
  6MWT
Changes in mMRC Dyspnoe Scale | 6 and 12 months
  mMRC

OTHER OUTCOMES:
Number and type of device-related and procedure-related serious adverse events (SAE) attributed to the use of RePneu LVRC | up to 6 months
  SAE device and procedure related

CONTACTS AND LOCATIONS:
Locations (2):
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark
- University Hospital of Saarland, Homburg, Saarland, Germany